CLINICAL TRIAL: NCT00858260
Title: Genetic Determinants of Phosphocalcic Metabolism in Hemodialysis Patients
Brief Title: Arnogene: A Phosphocalcic Study in Dialysis
Acronym: ARNOGENE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Pr Denis FOUQUE, Hospices Civils de Lyon
Other Study IDs: 2007.471/14
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Dialysis
Keywords: Klotho; calcium; phosphate; parathormone; survival; dialysis; Adult patients undergoing maintenance dialysis since at leat three months
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Searching for high morbi-mortality risk Klotho variants
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hemodialysis patients: Adult patients undergoing maintenance dialysis since at leat three months
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample — Searching for Klotho variants in DNA

SUMMARY:
Searching for high morbi-mortality risk Klotho variants in dialysis patients

ELIGIBILITY:
Inclusion Criteria:

* Every adult > 18 years old and treated by dialysis in centers located in the Rhone Alpes area in France.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing maintenance dialysis since at leat three months
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2008-11; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Assessing morbi-mortality based on Klotho variants

SECONDARY OUTCOMES:
Survival and serum phosphocalcic parameters

CONTACTS AND LOCATIONS:
Overall Officials: FOUQUE Denis, MD, Principal Investigator — Hospices Civils de Lyon; LEGRAND Eric, MD, Principal Investigator — CH Annonay; KAARASLAN Huseyin, MD, Principal Investigator — CH Bourgoin Jallieu; ABOKASEM Ayman, MD, Principal Investigator — CH Chalon/saône; LATAILLADE Claire Dominique, MD, Principal Investigator — CH Sallanches; KUENTZ François, MD, Principal Investigator — Centre Dialyse eaux claires; HACHACHE Toufic, MD, Principal Investigator — CHU Grenoble - La Tronche; LEITIENNE Philippe, MD, Principal Investigator — Hospices Civils de Lyon; ARKOUCHE Walid, MD, Principal Investigator — AURAL - Lyon; HEYANI Ahmed, MD, Principal Investigator — CH MACON; HANNOUN Jacques, MD, Principal Investigator — CH Villefranche/saône; COMBARNOUS François, MD, Principal Investigator — Clinique du Tonkin VILLEURBANNE; MAUREAUGANDRY Xavier, MD, Principal Investigator — AGDUC - Montélimar; SIRAJEDINE Mohamed, MD, Principal Investigator — CH ROMANS/ISERE; JEAN Ahmed, MD, Principal Investigator — Centre du Rein - Tassin la demi lune; DENICOLA Cora, MD, Principal Investigator — Calydial - CH Viennes
Locations (1):
- Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Derived] Marcais C, Maucort-Boulch D, Drai J, Dantony E, Carlier MC, Blond E, Genet L, Kuentz F, Lataillade D, Legrand E, Moreau-Gaudry X, Jean G, Fouque D; ARNOGENE Project. Circulating Klotho Associates With Cardiovascular Morbidity and Mortality During Hemodialysis. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3154-3161. doi: 10.1210/jc.2017-00104. PMID 28402487